CLINICAL TRIAL: NCT04955470
Title: Ketamine Infusion for Rapid Reduction of Suicidality in Pediatrics: a Pilot Randomized Controlled Trial
Brief Title: Ketamine Infusion for Rapid Reduction of Suicidality in Pediatrics
Acronym: Keta4SI
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: There were challenges with recruitment in the ED due to ED staffing shortages and we were unable to meet the expected recruitment rate. The decision to stop study recruitment was solely due to operational and logistical limitations.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Quynh Doan, Pediatric Emergency Physician and Associate Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H21-01433
Record Dates: First submitted 2021-06-21; First posted 2021-07-08 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Suicidal Ideation
MeSH Terms: conditions — Suicidal Ideation | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intravenous ketamine (Experimental): Infusion of 0.5 mg/kg of ketamine, at maximum dose of 40 mg, over 40 minutes.
  Interventions: Drug: Ketamine Injectable Solution
- Intravenous midazolam (Active Comparator): Infusion of 0.03 mg/kg of midazolam, at maximum dose of 2 mg, over 40 minutes.
  Interventions: Drug: Midazolam Injectable Solution
- Intravenous saline (Placebo Comparator): Infusion of 0.9% saline over 40 minutes.
  Interventions: Drug: Normal Saline 0.9% Injectable Solution

INTERVENTIONS:
Drug: Ketamine Injectable Solution — A 10 mg/mL solution of ketamine will be infused over a 40 minute period at a dose of 0.05mg/kg.
  Arms: Intravenous ketamine
Drug: Midazolam Injectable Solution — A 5 mg/mL solution of midazolam will be infused over a 40 minute period at a dose of 0.02 mg/kg.
  Arms: Intravenous midazolam
Drug: Normal Saline 0.9% Injectable Solution — A 0.9% normal saline solution will be infused over a 40 minute period.
  Arms: Intravenous saline

SUMMARY:
Suicide is a leading cause of death for children and adolescents. Since warning signs of suicide and links to precipitating events differ between age groups, suicide can be difficult to predict. As a result, children often seek care for suicidal ideation (SI) in the emergency department (ED) where a limited number of treatment options exist. Current psychotherapies and pharmacotherapies, such as antidepressants, provide benefit over weeks or months and thus limits their effective application in the ED. Consequently, when there is an imminent threat to the child's safety, the typical management solution is to admit the patient to a safe environment and hopefully de-escalate over time. To address a more rapid-onset treatment option for SI, a number of studies in adults have suggested that a single, sub-anesthetic dose of intravenous ketamine can rapidly reduce depression and SI severity. These results are promising, but large-scale trials are needed to determine if ketamine is a safe and effective treatment for acute suicidality in the pediatric population. This approach has the benefit of working rapidly, avoiding involuntary hospitalizations, and protecting patients from self-harm until they can be connected to longer term mental health resources. This study will compare the use of intravenous ketamine to both active and placebo controls in children 10 to 17 years of age presenting to the pediatric ED for SI. The primary objective of this pilot trial is to explore the adequacy and range of three instruments measuring suicidality and to determine the sample size required for a large definitive randomized control trial. This larger trial will be used to estimate the effectiveness of intravenous ketamine for reducing SI in children in the pediatric ED. The secondary objectives are to assess study feasibility and optimize study procedures. Given very few side effects reported in adult studies and the relatively benign nature of those reported, the investigators do not expect any major safety concerns in the study.

ELIGIBILITY:
The study will enroll children and adolescents presenting with SI in the paediatric ED.

Inclusion Criteria:

1. 10 to 17 years of age
2. Respond "yes" to either question 1 (Passive Ideation) or 2 (Active Ideation) on the C-SSRS
3. Respond "yes" to either questions 3 (Method), 4 (Intent), or 5 (Plan) on the C-SSRS
4. Deemed acceptable and appropriate for admission to the on-site Child and Adolescent Psychiatry Emergency (CAPE) unit by a pediatric psychiatrist
5. Successful completion of Capacity to Assent.
6. Normal vital signs for age and a normal neurological exam (no focal deficits or abnormalities), as per attending clinician

Exclusion Criteria:

1. History of benzodiazepine or ketamine use in the past 3 months (ample wash out period)
2. Lifetime history of ketamine or benzodiazepine use disorder
3. Previous diagnosis of schizophrenia or active psychosis as per the treating physician
4. Lifetime history of schizoaffective disorder
5. Current hypomania, mania, mixed state
6. Clinically unstable, requires resuscitation or admission to a medical ward for stabilizing therapy (i.e., intensive care unit.)
7. History of cerebrovascular accident, uncontrolled seizure disorder, increased intracranial pressure
8. Uncontrolled hypertension, low or labile blood pressure, severe cardiac decompensation
9. Moderate to severe hepatic/renal impairment
10. Intoxicated or delirious
11. Suspected or confirmed pregnancy or women who are breastfeeding
12. Known allergy or sensitivity to ketamine and/or midazolam or any component in the formulation.
13. Neuro-cognitive impairment that precludes informed consent, assent, or ability to self-report pain and satisfaction
14. Inability to understand spoken and/or written English without the use of an interpreter
15. Previous enrollment in this study
16. No parent/guardian present.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) | 90 minutes post infusion
  The CSSR-S is 6-point scale that measures SI severity via clinical interviews, ranging from 1 (wish to be dead) to 5 (suicidal intent with plan). Adolescents who deny any SI receive a 0. The distribution of "yes" responses on questions 3, 4, or 5 will be assessed from baseline. Higher scores indicate greater SI severity.
Montgomery-Åsberg Depression Rating Scale (MADRS) | 90 minutes post infusion
  The MADRS is a 10-item, 6-point scale that screens for depressive symptoms in adults via clinical interviews. A self-reported version (MADRS-self assessment) which has been validated in adolescents will be used, but only the final item that is specific to SI (item 10) will be asked. The distribution of scores from 0 to 6 will be assessed from baseline. Higher scores indicate greater SI severity.
Pragmatic questionnaire | 90 minutes post infusion
  The pragmatic questionnaire is a brief, one sentence question designed to assess change in SI. Participants will be asked "How suicidal do you feel on a scale of 0 to 10?". The distribution of scores from 0 to 10 will be assessed from baseline. Higher scores indicate greater SI severity.

SECONDARY OUTCOMES:
Columbia Suicide Severity Rating Scale (C-SSRS) | 24 hours
  The CSSR-S is 6-point scale that measures SI severity via clinical interviews, ranging from 1 (wish to be dead) to 5 (suicidal intent with plan). Adolescents who deny any SI receive a 0. The distribution of "yes" responses on questions 3, 4, or 5 will be assessed from baseline. Higher scores indicate greater SI severity.
Montgomery-Åsberg Depression Rating Scale (MADRS) | 24 hours, 7-, 14-, 21-, and 28 days
  The MADRS is a 10-item, 6-point scale that screens for depressive symptoms in adults via clinical interviews. A self-reported version (MADRS-self assessment) which has been validated in adolescents will be used, but only the final item that is specific to SI (item 10) will be asked. The distribution of scores from 0 to 6 will be assessed from baseline. Higher scores indicate greater SI severity.
Pragmatic questionnaire | 24 hours, 7-, 14-, 21-, and 28 days
  The pragmatic questionnaire is a brief, one sentence question designed to assess change in SI. Participants will be asked "How suicidal do you feel on a scale of 0 to 10?". The distribution of scores from 0 to 10 will be assessed from baseline. Higher scores indicate greater SI severity.
Blinding assessment | 90 minutes post infusion
  The proportion of participants and research personnel that correctly identify treatment arm allocation.
Enrolment rate | 28-days
  Proportion of eligible patients that consent to participate, and proportion of participants that are lost to follow-up at 7-, 14-, 21-, and 28-days.
Demographics | 28-days
  Demographics of eligible patients who decline to participate in the study.
Drug reactions | 28-days
  Incidence and frequency of side effects and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh Doan, PhD MHSc MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No